CLINICAL TRIAL: NCT03582280
Title: Study to Improve the Function and Welfare of Late-stage Solid Cancer Subjects by Amorphous Calcium Carbonate (ACC) Treatment, Administered Orally and Concomitantly With Inhalation
Brief Title: The Effect of Amorphous Calcium Carbonate (ACC) Treatment on Function and Welfare in Late-stage Solid Cancer Subjects
Acronym: ONCO-004-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCS-ONCO-004-1
Record Dates: First submitted 2018-06-19; First posted 2018-07-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amorous Calcium Carbonate (ACC) - Amor (Experimental): The investigational product will include:
  1. Amor powder, each eppendorf contains 200mg Calcium
  2. Amor Inhaled Double Pack - 1% ACC in 8 ml suspension
  Interventions: Drug: Amorphous Calcium Carbonate (ACC) - Amor

INTERVENTIONS:
Drug: Amorphous Calcium Carbonate (ACC) - Amor — Amor Powder is composed of Amorphous Calcium Carbonate and is administered oral Amor Inhaled Double Pack is composed of 1% ACC in solution and is administered by inhalation

SUMMARY:
An exploratory open label study to improve the function and welfare of late-stage solid cancer subjects (with or without lung involvement) who failed or refused anti-cancer treatment by ACC treatment, administered orally and concomitantly by inhalation.

The following measures will be evaluated: improvement of pain, performance status, dyspnea measurement (Modified Borg Scale)/ oxygen saturation (if applicable) and overall survival.

The subjects' medical charts will be reviewed for their eligibility including the following: medical history, prior cancer treatments, pathologic diagnosis of cancer, and CT/Chest X-ray results. Assessment of prior and concurrent medication use, physician evaluation of patient status, and measurement of Albumin Corrected Serum Calcium level (to be done at baseline and prior to dose escalation, so that results are available prior to the visit) will be performed prior to each dose escalation; in addition, vital signs, ECOG/Karnofsky performance status and VAS pain assessments will be recorded at each visit as well. CT test will be executed during the study period: at baseline, week 12 and week 24 visits in order to assess progression free survival by CT.

The tests during the visits will be performed by a physician/nurse. Each subject will receive individual doses of AMOR-powder by escalating doses up to 1,800 mg of ACC powder per day (Amor powder administration will be continuous along the day - each eppendorf every two hours). Patients who will not be able to swallow the powder, will receive similar doses of ACC in tablets.

In addition, subject will inhale 1% ACC in 8 ml suspension, for inhalation three times a day.

Subject's functionality will be assessed by serially determining ECOG/Karnofsky performance status. Subject's progression free survival will be assessed by CT to evaluate tumor response to treatment.

DETAILED DESCRIPTION:
Subjects diagnosed with late stage solid cancer (with or without lung involvement) who failed or refused anti-cancer treatment will be enrolled and administered with both: AMOR powder up to 1800 mg daily and AMOR Inhaled Double Pack 1% ACC in 8 ml suspension - three times a day.

Starting Doses:

1200 mg of AMOR powder (will be administered continuously along the day, each Eppendorf every two hours) scaled up by 200 mg every week until maximum dose of 1,800 mg. Patients who will not be able to swallow the powder, will receive similar doses of ACC tablets.

ACC Amor Inhaled Double Pack; 1% ACC in 8 ml suspension - for inhalation three times a day.

Screening hospital visit:

* Inform consent
* Subjects' medical charts will be reviewed for medical history, prior cancer treatments
* Eligibility Criteria assessment: adherence with inclusion/exclusion criteria
* Pathologic diagnosis of cancer and CT/Chest X-Ray will be obtained from the patient's charts as needed.
* Concomitant medications
* Physician evaluation of patient status
* Lab: Hematology, Blood chemistry, Albumin Corrected Serum Calcium will be performed prior to first dose (blood to be drawn in the morning before breakfast)
* Serum 25-hydroxy-vitamin D, i.e. 25(OH)D
* Pain VAS score scale
* ECOG/Karnofsky performance status
* Vital signs (blood pressure and heart rate - supine, respiration rate (RR), oral body temperature)
* Weight
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* All women of child-bearing potential will have a pregnancy test
* Once eligibility criteria are met, subject will undergo CT imaging during screening or baseline or week 1 visit.
* Following CT, RECIST ver. 1.1 Once eligibility criteria are met, subject will initiate treatment of ACC. Vitamin D levels will be re-examined and recorded.

Baseline (Week 0) hospital visit:

* Eligibility Criteria assessment: adherence with inclusion/exclusion criteria
* Subjects' medical charts will be reviewed for medical history, prior cancer treatments
* Concomitant medications
* Lab: Hematology, Blood chemistry, Albumin Corrected Serum Calcium will be performed prior to first dose (blood to be drawn in the morning before breakfast; must have calcium level measurement before escalation)
* Serum 25-hydroxy-vitamin D, i.e. 25(OH)D
* VAS once daily
* ECOG/Karnofsky performance status
* Vital signs (blood pressure and heart rate - supine, respiration rate (RR), oral body temperature)
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* All women of child-bearing potential will have a pregnancy test
* CT imaging to evaluate tumor size and volume at study initiation, if test was not performed between the screening and baseline visit.
* RECIST ver. 1.1 (if was not performed during screening visit).

First ACC Dose:

* ACC Per Os (PO) 1200 mg x1 (i.e. 6 AMOR powder Eppendorf's daily, (Amor powder administration will be continuous along the day, i.e. each Eppendorf will be administered every two hours). Patients who will not be able to swallow the powder, will receive similar doses of ACC tablets.
* ACC 1% in 8 mL suspension- inhalation for three times a day.

Week 1 (+/- 2 days range) hospital visit:

* Albumin Corrected Serum Calcium will be performed prior to dose escalation (blood to be draw in the morning before breakfast)
* Dose escalation of ACC PO by 200 mg for a total daily dose of 1400 mg (Amor powder administration will be continuous along the day)
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* VAS once daily
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* CT imaging to evaluate tumor size and volume at study initiation, if test was not performed during screening visit.
* RECIST ver. 1.1 (if was not performed during baseline visit).
* AEs/DLTs

Week 2 (+/- 2 days range) hospital visit:

* Albumin Corrected Serum Calcium will be performed prior to dose escalation (blood to be draw in the morning before breakfast)
* Dose escalation of ACC PO by 200 mg for a total daily dose of 1600 mg (Amor powder continuous administration along the day)
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* VAS once daily
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* AEs/DLTs

Week 3 (+/- 2 days range) hospital visit/ home visit:

* Albumin Corrected Serum Calcium will be performed prior to dose escalation (blood to be draw in the morning before breakfast)
* Dose escalation of ACC PO by 200 mg for a total daily dose 1800 mg (Amor powder administration will be continuous along the day)
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* VAS once daily
* ECOG/Karnofsky performance status
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* AEs/DLTs

Treatment Maintenance:

Week 6 (+/- 2 days range) hospital visit:

* ACC PO administration will be continuous along the day at the final patient dosage level
* Albumin Corrected Serum Calcium
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* Physician evaluation of patient status
* Hematology
* Blood chemistry
* ECOG/Karnofsky performance status
* Pain VAS scale score
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* AEs/DLTs

Week 12 (+/- 2 days range) hospital visit:

* ACC PO administration will be continuous along the day at the final patient dosage level
* Albumin Corrected Serum Calcium
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* Physician evaluation of patient status
* Hematology
* Blood chemistry
* CT imaging to evaluate tumor size and volume
* RECIST ver. 1.1
* ECOG/Karnofsky performance status
* Pain VAS scale score
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* AEs/DLTs

Week 18 (+/- 2 days range) hospital visit:

* ACC PO administration will be continuous along the day at the final patient dosage level
* Albumin Corrected Serum Calcium
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* Physician evaluation of patient status
* Hematology
* Blood chemistry
* ECOG/Karnofsky performance status
* Pain VAS scale score
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* AEs/DLTs

Week 24 Termination visit (+/- 2 days range) hospital visit:

* ACC PO administration will be continuous along the day at the final patient dosage level
* Albumin Corrected Serum Calcium
* ACC 1% in 8 mL suspension- inhalation for three times a day.
* Concomitant medications
* Physician evaluation of patient status
* Hematology
* Blood chemistry
* CT imaging to evaluate tumor size and volume at study endpoint
* RECIST ver. 1.1
* ECOG/Karnofsky performance status
* Pain VAS scale score
* Oxygen saturation as determined by pulse oximeter/ Dyspnea measurement (Modified Borg Scale)
* AEs/DLTs A decision regarding a follow up period will be made at the discretion of the investigator based on the subject's condition together with subject's agreement. Once agree, study drugs will be dispensed for the follow up period. The follow up period will be prolonged up to 6 months following study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 18 years +
2. Signed the informed consent
3. Late Stage Histologically proven advanced solid tumours for which no standard of care therapy exist or failed or refused anti-cancer treatment
4. Subject should not have any illness or condition deemed by the physician to contra-indicate treatment with ACC or may interfere with the assessment of the therapy
5. Performance Status: ECOG 0-3/ Karnofsky performance status >50
6. Life Expectancy : at least 2 months
7. Hormonal therapy is allowed if needed
8. Patient is on conservative treatment for relieving his symptoms
9. Subjects within normal range of serum-corrected albumin calcium (between 7.0-10.5 mg/dl)
10. Acceptable haematology and biochemistry variables:

    WBC ≥3000/mm3 Absolute Neutrophil count ≥ 1500 /mm3 Platelet Count ≥ 100,000/mm3 Hemoglobin ≥ 9 g/dL Bilirubin ≤ 1.5 x ULN ALT and AST ≤ 2.5 x ULN; for patients with hepatic metastases, ALT and AST ≤ 5 x ULN PT/PTT ≤ 1.5 ULN
11. Subjects should have sufficient Vitamin D levels upon study entry, which is defined as 25(OH)D serum level >20 ng/mL (50 nmol/L) according to a document composed by the Food and Nutrition Board of the Institute of Medicine, USA. If the subject is Vitamin D insufficient or deficient, then a loading dose of Vitamin D3 will be administered during subject's enrollment or during the study as follows:

    1. If the serum 25(OH)D level is 12-20 ng/mL (30-50 nmol/L) then a loading oral dose of 50,000 IU of Vitamin D3 should be administered twice with 3-5 days in between the doses.
    2. If the serum 25(OH)D level is ≤ 12 ng/mL (30 nmol/L), then a loading oral dose of 50,000 IU of Vitamin D3 will be administered three times with 3-5 days in between the doses. Serum 25(OH)D levels will be checked 1-2 weeks following the last loading.
12. Subjects receiving Denosumab or bisphosphonates are eligible. Denosumab or bisphosphonates can be administered during the study to alleviate bone metastasis pain.
13. Negative Pregnancy Test.

Exclusion Criteria:

1. Concurrent treatment with acute anti-cancer therapy
2. Hypercalcemia or previous consistent reporting of hypercalcemia (serum calcium concentration > 12.0 mg/dL)
3. Clinical Significant Cardiovascular Disease
4. Known alcohol or drug abuse
5. Any psychiatric condition that would prohibit understanding or rendering of Informed Consent
6. Active Participation in Clinical Trial in the last 2 weeks prior to inclusion
7. Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment.
8. Nephrolithiasis
9. Pregnancy

   -

Ages: 18 Years to 119 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) score for pain | week 0, week 1, week 2, week 3, week 6, week 12, week 18, week 24
  Assessing a change in Pain VAS score The scale is between 0-10. 0 is a score for no pain 5 is a score for moderate pain 10 is a score for unbearable pain
ECOG Performance status (PS) | week 0, week 1, week 2, week 3, week 6, week 12, week 18, week 24
  Assessing a change in PS Grade 0 - Fully active, able to carry on all pre-disease performance without restriction Grade1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work Grade 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours Grade 3 - Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours Grade 4 - Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair Grade 5 - Dead
Oxygen saturation | week 0, week 1, week 2, week 3, week 6, week 12, week 18, week 24
  Assessing a change in oxygen saturation Normal pulse oximeter readings usually range from 95 to 100 percent. Values under 90 percent are considered low.
Progression Free Survival | week 0, week 12, week 24
  Assessing a change from baseline in tumor's growth and size by using CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Carem, Jerusalem, Israel